CLINICAL TRIAL: NCT00539396
Title: A Phase 2 Randomized, Open Label, Multi-Center Study of the Use of Prandial Inhaled Technosphere Insulin in Combination With Basal Subcutaneous Lantus as Basal Insulin Versus Prandial Subcutaneous NovoRapid in Combination With Basal Subcutaneous Lantus Insulin in Subjects With Type 1 Diabetes Mellitus
Brief Title: A 3 Month, Randomized, Open Label, Multi-center Study of Technosphere/Insulin Compared to Insulin Aspart in Subjects With Type 1 Diabetes Mellitus Receiving Insulin Glargine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-101
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Technosphere Insulin

SUMMARY:
A 3 month, randomized, open label, multi-center study of Technosphere/Insulin compared to insulin aspart in subjects with type 1 diabetes mellitus receiving insulin glargine

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes currently receiving SC insulin at mealtimes for at least 3 months
* BMI <40 kg/m squared
* HbA1c greater than or equal to 7% and less than or equal to 11.5%
* Serum creatinine less than 2 for males and less than 1.8 for females
* Acceptable pulmonary function

Exclusion Criteria:

* Significant hepatic disease
* Previously diagnosed pulmonary disease, ketoacidosis of evidence of severe secondary complications of diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2005-03; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose following a standard meal | 0-300 minutes

SECONDARY OUTCOMES:
Mean change from baseline HbA1c | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Robert Baughman, PhD, Study Director — Mannkind Corporation